CLINICAL TRIAL: NCT04304469
Title: Management of Women Who Experience Domestic Abuse: a Feasibility Study Comparing Psychological Outcomes at the Maison Des Femmes in Saint-Denis and a Convential Shelter
Brief Title: Management of Women Who Experience Domestic Abuse: Study Comparing Psychological Outcomes at the Maison Des Femmes in Saint-Denis and a Convential Shelter
Acronym: AVEC-L
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BARDOU THELLIE 2019
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Domestic Violence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women: women consulting for domestic violence
  Interventions: Other: surveys; Other: follow-up

INTERVENTIONS:
Other: surveys — delivery of the survey at a domestic violence consultation
Other: follow-up — follow-up of women 6 months after their consultation

SUMMARY:
ach year, it is estimated that an average of approximately 219,000 women in France suffer physical and/or sexual violence at the hands of their partner or ex-partner. These figures do not take into account other types of violence such as psychological or economic violence. Domestic violence has a major impact on the physical, sexual and psychological health of women victims. For example, the prevalence of post-traumatic stress disorder in these women varies between 33 and 84%, with an average prevalence of 61%, compared with only 2.2% in the French population as a whole. Multidisciplinary medical, social and legal support for these women is essential. In France, there are major territorial disparities in terms of the distribution of facilities for victims of domestoc violence, and not all women victims have the same access to care depending on their place of residence.

The Maison des Femmes in St Denis has been open since 2016. It offers a unique range of sanitary, social and judicial services through cooperation with police and justice departments, for women who have been subjected to any type of violence.

This facility is unique in France, and the number of consultations continues to increase, and was more than 8,500 in 2018. The Maison des Femmes model is intended to be exported to other departments, but first the model needs to be validated, beyond its obvious attractiveness (illustrated by the number of consultations and the fact that it attracts women from throughout the Ile de France region) by comparing it to other facilities in terms of its effect on the management of the women.

This is a cross-sectional prevalence study that estimates the frequency of post-traumatic stress disorder among women who are victims of domestic violence who used the services offered at the Maison des Femmes or other dedicated structures, at the initial consultation and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 and over,
* Consulted for domestic violence at the Maison des Femmes, St Denis health centre or Aubervilliers health centre.
* Able to understand the objectives of the study and to respond to the survey
* Having been informed and not having objected to participating in this study.

Exclusion Criteria:

* Unable to understand the objectives of the study and to respond to the surveys.
* Consulting for another reason.
* Protected adult under a measure of safeguard.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women consulting for domestic violence
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Prevalence of Post-Traumatic Stress Disorder by PCL-5 Scale | at the end of study, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Roland N, Delmas N, El Khoury F, Bardou A, Yacini L, Feldmann L, Hatem G, Mahdjoub S, Bardou M. Post-traumatic stress disorders in women victims-survivors of intimate partner violence: a mixed-methods pilot study in a French coordinated structure. BMJ Open. 2024 Jan 23;14(1):e075552. doi: 10.1136/bmjopen-2023-075552. PMID 38262657